CLINICAL TRIAL: NCT04668391
Title: Ultrasound-guided Anterior Quadratus Lumborum Block at the Lateral Supra-arcuate Ligament Versus Thoracic Epidural Analgesia After Open Liver Surgery: A Prospective, Randomized, Controlled, Noninferiority Trial
Brief Title: Anterior Quadratus Lumborum Block at the Lateral Supra-arcuate Ligament for Analgesia After Open Liver Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, Huifang Jiang, Principal Investigator, Zhejiang Cancer Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-2020-350
Record Dates: First submitted 2020-12-13; First posted 2020-12-16 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-06

CONDITIONS: Liver Surgery
MeSH Terms: interventions — Tea

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Quadratus lumborum block (Experimental): Ultrasound-guided anterior quadratus lumborum block at the lateral supra-arcuate ligament.
  Interventions: Procedure: Ultrasound-guided anterior quadratus lumborum block at the lateral supra-arcuate ligament
- Thoracic epidural analgesia (Active Comparator): Thoracic epidural analgesia at the level of T7-10.
  Interventions: Procedure: Thoracic epidural analgesia

INTERVENTIONS:
Procedure: Ultrasound-guided anterior quadratus lumborum block at the lateral supra-arcuate ligament — Bilateral single-injection 20 ml 0.56% ropivacaine. Intravenous analgesia was started postoperatively and consisted of 1ug/ml sufentanil，2 ml/h with a 5-minute lockout period, a limited 12 ml/h dose.
  Arms: Quadratus lumborum block
Procedure: Thoracic epidural analgesia — A thoracic epidural at the level of T7-10. Epidural infusion was started postoperatively and consisted of sufentanil (0.6ug/mL) and ropivacaine（0.2%） at 3ml/h.
  Arms: Thoracic epidural analgesia

SUMMARY:
This is a prospective, randomized, controlled, noninferiority trial for evaluating the efficacy of ultrasound-guided anterior quadratus lumborum block at the lateral supra-arcuate ligament versus thoracic epidural analgesia after open liver surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age≥18 years
* ASA I-III
* Open liver surgery

Exclusion Criteria:

* Contraindication to nerve block or epidural puncture
* Chronic use of opioids or NSAIDs
* Refused to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2020-12-17 (Actual); Primary Completion 2021-06-02 (Actual); Study Completion 2021-07-02 (Actual)

PRIMARY OUTCOMES:
NRS (numeric rating scale) score for coughing pain | at 24 hours after surgery
  Postoperative pain was assessed by NRS score with a range of 0 to 10 (0=no pain, 10=the worst possible pain)

SECONDARY OUTCOMES:
NRS score for rest and coughing pain | at 1, 6, 24, 48, 72 hours after surgery
  Postoperative pain at rest and during coughing was assessed by NRS score with a range of 0 to 10 (0=no pain, 10=the worst possible pain)
consumption of opioid converted to IV morphine equivalents | during 24 hours after surgery
  opioids given postoperatively converted to IV morphine equivalents
Numbers of additional analgesics | during 72 hours after surgery
  Additional rescue analgesics were used when pain relief was inadequate (NRS >3). The choice of rescue analgesic was oxydone 5-10mg.
The incidence of postoperative hypotension | during 72 hours after surgery
  Adverse reactions related to analgesia
The incidence of nausea and vomiting | during 72 hours after surgery
  Adverse reactions related to analgesia
The incidence of pruritus | during 72 hours after surgery
  Adverse reactions related to analgesia
The incidence of respiratory depression | during 72 hours after surgery
  Adverse reactions related to analgesia
Time to ambulation in days | through study completion, an average of 2-3 days
  Postoperative ambulation time
Time to eat in days | through study completion, an average of 2-3 days
  Time to start eating after surgery
Time to flatus in hours | through study completion, an average of 40-50 hours
  Time to flatus after surgery
Time to defecation in hours | through study completion, an average of 60-70 hours
  Time to defecation after surgery
Time to urethral catheter removal in hours | through study completion, an average of 60-70 hours
  Time tourethral catheter removal after surgery
Postoperative hospital stay in days | through study completion, an average of 7-8 days
  The time from operation to discharge
Clavien-Dindo classification (grade I, II, III, IV) for postoperative complication | One month after surgery
  Postoperative Clavien-Dindo complication classification

CONTACTS AND LOCATIONS:
Overall Officials: Huifang Jiang, M.D., Principal Investigator — Zhejiang Caner Hospital
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Yes
Postoperative numeric rating scale (NRS) pain score at rest and during coughing at 1, 6, 24, 48 and 72 hours after surgery.
Time Frame: permanent validity
Access Criteria: Baidu Netdisk code：3i81
URL: http://pan.baidu.com/s/1EZkWQ6GkhoNBaWCJhUd1PA

REFERENCES:
- [Background] Li H, Ma D, Liu Y, Wang Y. A transverse approach for ultrasound-guided anterior quadratus lumborum block at the lateral supra-arcuate ligament. Anaesthesia. 2020 Oct;75(10):1400-1401. doi: 10.1111/anae.15058. Epub 2020 Jun 24. No abstract available. PMID 32578192
- [Derived] Gu B, Zhou H, Lian Y, Zhou Y, He S, Xie K, Jiang H. Ultrasound-Guided Anterior Quadratus Lumborum Block at Lateral Supra-Arcuate Ligament vs Thoracic Epidural Analgesia after Open Liver Surgery: A Randomized, Controlled, Noninferiority Trial. J Am Coll Surg. 2022 Dec 1;235(6):871-878. doi: 10.1097/XCS.0000000000000354. Epub 2022 Nov 15. PMID 36102582